CLINICAL TRIAL: NCT02712359
Title: Long Term Hepatitis A Virus (HAV) Antibody Persistence in Children Vaccinated With 1 Dose and Those Vaccinated With 2 Doses of Havrix in Panama
Brief Title: This Study Will Evaluate the Persistence of Hepatitis A Antibodies, 8 Years and 10 Years Later, in Children Who Had Received Havrix at Selected Health Centres of Panama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201630
Record Dates: First submitted 2016-03-07; First posted 2016-03-18 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis A Vaccine
Keywords: Havrix; Cross-sectional seroprevalence survey; Panama; Long-term persistence; Hepatitis
MeSH Terms: conditions — Hepatitis

ARMS (4):
- Havrix 1 dose_Year 8 Group (Other): Subjects who received one dose of Havrix vaccine and with more than or equal to (≥) 7 years and less than (<) 10 years between the administration of the vaccine dose and the Persistence Visit at Year 8 and who participated in the Year 8 cross-sectional survey.
  Interventions: Other: Blood sample collection
- Havrix 2 doses_Year 8 Group (Other): Subjects who received two doses of Havrix vaccine and with more than or equal to (≥) 7 years and less than (<) 10 years between the administration of the last vaccine dose and the Persistence Visit at Year 8 and who participated in the Year 8 cross-sectional survey.
  Interventions: Other: Blood sample collection
- Havrix 1 dose_Year 10 Group (Other): Subjects who received one dose of Havrix vaccine and with more than or equal to (≥) 10 years and less than (<) 13 years between the administration of the vaccine dose and the Persistence Visit at Year 10 and who participated in the Year 10 cross-sectional survey.
  Interventions: Other: Blood sample collection
- Havrix 2 doses_Year 10 Group (Other): Subjects who received two doses of Havrix vaccine and with more than or equal to (≥) 10 years and less than (<) 13 years between the administration of the vaccine dose and the Persistence Visit at Year 10 and who participated in the Year 10 cross-sectional survey.
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — A blood sample (~5mL) will be collected from all subjects at each cross-sectional survey (Year 8 and Year 10).

SUMMARY:
The purpose of this study is to evaluate the persistence of hepatitis A antibodies, approximately 8 years and 10 years post vaccination with the complete series of Havrix (2 doses) and the partial series completion (1 dose).

DETAILED DESCRIPTION:
The study comprises of two independent cross-sectional surveys (Year 8 and Year 10). The first cross-sectional serosurvey will evaluate the long term persistence of immunity approximately 8 years post vaccine administration and the second cross-sectional study will evaluate long term persistence, approximately 10 years post vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parent(s)/ LAR(s), in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed assent/consent obtained from the subject or subject's parent(s)/ LAR(s) of the subject.
* Available HAV vaccination records.
* Children who have received either 1 or two doses of Havrix at selected health centres of Panama.
* Children with ≥ 7 years and < 10 years between last dose and Persistence Visit 1 (Year 8) and children ≥ 10 years and < 13 years between last dose and Persistence Visit 1' (Year 10).

Exclusion Criteria:

* Child in care.
* Subjects with history of vaccination with other hepatitis A vaccines other than Havrix.
* Subjects with known past history of hepatitis A infection, both without vaccination and after they received the last dose of Havrix (1 dose or the complete 2 dose schedule).

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1201 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Panama (3):
  - GSK Investigational Site, Chiriquí
  - GSK Investigational Site, Juán Diaz
  - GSK Investigational Site, Panama City

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in Panama. Out of the 1201 subjects originally enrolled in the study, 2 subjects were eliminated from the ATP cohort for persistence, due to non-eligibility. Hence, 1199 subjects were included in the ATP cohort for persistence.
Pre-assignment Details: The design of the study included 2 epochs: Epoch 001 - Persistence at Year 8 and Epoch 002 - Persistence at Year 10.
Period: Epoch 001: Persistence at Year 8
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group
Started | 300 | 300 | 0 | 0
Completed | 300 | 300 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Epoch 002: Persistence at Year 10
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group
Started | 0 | 0 | 299 | 300
Completed | 0 | 0 | 299 | 300
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The demographic characteristics are presented separately for each study epoch (Epoch 001: Persistence at Year 8 and Epoch 002: Persistence at Year 10).
Groups:
- Total: Total of all reporting groups
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group | Total
Number analyzed (Participants) | 300 | 300 | 299 | 300 | 1199
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age continuous data for Epoch 001: Persistence at Year 8 Population: The age continuous data in this baseline measure are reported for Havrix 1 dose_Year 8 and Havrix 2 doses_Year 8 Groups.
  Years
    number analyzed (Participants) | 300 | 300 | 0 | 0 | 600
    (all) | 10.5 (0.9) | 10.0 (0.7) |  |  | 10.2 (0.8)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age continuous data for Epoch 002: Persistence at Year 10 Population: The age continuous data in this baseline measure are reported for Havrix 1 dose_Year 10 and Havrix 2 doses_Year 10 Groups.
  Years
    number analyzed (Participants) | 0 | 0 | 299 | 300 | 599
    (all) |  |  | 12.0 (0.5) | 12.0 (0.4) | 12.0 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex: Female, Male data for Epoch 001: Persistence at Year 8 Population: The sex: female, male data in this baseline measure are reported for Havrix 1 dose_Year 8 and Havrix 2 doses_Year 8 Groups.
  Participants
    number analyzed (Participants) | 300 | 300 | 0 | 0 | 600
    Female | 136 | 160 | 0 | 0 | 296
    Male | 164 | 140 | 0 | 0 | 304
Sex: Female, Male [Count of Participants; unit: Participants] — Sex: female, male data for Epoch 002: Persistence at Year 10 Population: The sex: female, male data in this baseline measure are reported for Havrix 1 dose_Year 10 and Havrix 2 doses_Year 10 Groups.
  Participants
    number analyzed (Participants) | 0 | 0 | 299 | 300 | 599
    Female | 0 | 0 | 161 | 162 | 323
    Male | 0 | 0 | 138 | 138 | 276
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity data for Epoch 001: Persistence at Year 8 Population: The race/ethnicity data in this baseline measure are reported for Havrix 1 dose_Year 8 and Havrix 2 doses_Year 8 Groups.
  Participants
    Geographic Ancestry: number analyzed (Participants) | 300 | 300 | 0 | 0 | 600
    Geographic Ancestry: African Heritage / African American | 13 | 6 | 0 | 0 | 19
    Geographic Ancestry: White - Caucasian / European Heritage | 1 | 0 | 0 | 0 | 1
    Geographic Ancestry: Mixed Race | 286 | 294 | 0 | 0 | 580
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/ethnicity data for Epoch 002: Persistence at Year 10 Population: The race/ethnicity data in this baseline measure are reported for Havrix 1 dose_Year 10 and Havrix 2 doses_Year 10 Groups.
  Participants
    Geographic ancestry: number analyzed (Participants) | 0 | 0 | 299 | 300 | 599
    Geographic ancestry: African Heritage / African American | 0 | 0 | 5 | 6 | 11
    Geographic ancestry: American Indian or Alaskan Native | 0 | 0 | 3 | 1 | 4
    Geographic ancestry: White - Caucasian / European Heritage | 0 | 0 | 4 | 3 | 7
    Geographic ancestry: Mixed race | 0 | 0 | 287 | 290 | 577

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis A Virus (HAV) Seropositivity Status at Approximately 8 Years Following Last Administered Havrix Dose
Description: Subjects are defined as being seropositive if their anti-HAV antibody concentration is equal to or above (≥) 15 milli-international unit/milliliter (mIU/mL).
Time Frame: At approximately 8 years after the last administered vaccine dose
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for persistence at Year 8, which included all enrolled subjects who had a valid informed consent, had available assay results at Year 8 sero-surveys, had not received other HAV vaccine, with no history HAV infection prior to the study and who had available HAV vaccination records.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group
Number analyzed (Participants) | 300 | 300
Participants
  Seropositive | 223 | 293
  Seronegative | 77 | 7

2. Primary Outcome: Number of Subjects With Anti-HAV Seropositivity Status at Approximately 10 Years Following Last Administered Havrix Dose
Description: Subjects are defined as being seropositive if their anti-HAV antibody concentration is equal to or above (≥) 15 mIU/mL.
Time Frame: At approximately 10 years after the last administered vaccine dose
Population: The analysis was performed on the ATP cohort for persistence at Year 10, which included all enrolled subjects who had a valid informed consent, had available assay results at Year 10 sero-surveys, had not received other HAV vaccine, with no history HAV infection prior to the study and who had available HAV vaccination records.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group
Number analyzed (Participants) | 299 | 300
Participants
  Seropositive | 215 | 289
  Seronegative | 84 | 11

3. Secondary Outcome: Anti-HAV Antibody Concentrations at Approximately 8 Years Following Last Administered Havrix Dose
Description: Anti-HAV antibody concentrations were measured by ELISA, expressed as GMCs, in mIU/mL. The cut-off of the assay was an anti-HAV antibody concentration equal to or above (≥) 15 mIU/mL.
Time Frame: At approximately 8 years after the last administered vaccine dose
Population: The analysis was performed on the ATP cohort for persistence at Year 8, which included all enrolled subjects who had a valid informed consent, had available assay results at Year 8 sero-surveys, had not received other HAV vaccine, with no history HAV infection prior to the study and who had available HAV vaccination records.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group
Number analyzed (Participants) | 300 | 300
mIU/mL | 40.2 [34.2 to 47.4] | 123.9 [111.5 to 137.7]

4. Secondary Outcome: Anti-HAV Antibody Concentrations at Approximately 10 Years Following Last Administered Havrix Dose
Description: as for outcome 3
Time Frame: At approximately 10 years after the last administered vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group
Number analyzed (Participants) | 299 | 300
mIU/mL | 26.0 [23.0 to 29.5] | 82.1 [73.2 to 92.0]

5. Secondary Outcome: Number of Subjects With Anti-HAV Antibody Concentration ≥ 15 mIU/mL at Approximately 8 Years Following Last Administered Havrix Dose - Exploration of Non-inferiority of the 1-dose Schedule Compared to the 2-dose Schedule of Havrix
Description: Subjects are defined as being seropositive if their anti-HAV antibody concentration is equal to or above (≥) 15 mIU/mL.
Time Frame: At approximately 8 years after the last administered vaccine dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group
Number analyzed (Participants) | 300 | 300
Participants | 223 | 293
Statistical Analysis 1: Comparison: Havrix 1 dose_Year 8 Group vs Havrix 2 doses_Year 8 Group; Difference in seropositivity rates for anti-HAV antibody: To demonstrate that 1-dose schedule of Havrix (Havrix 1 dose_Year 8 Group) was non-inferior to the 2-dose schedule of Havrix (Havrix 2 doses_Year 8 Group), in terms of seropositivity rates for anti-HAV antibody, measured by ELISA, approximately 8 years after the administration of the last vaccine dose; Test type: Non-Inferiority — The lower limit of the 2-sided 95% confidence interval (CI) for the difference (Havrix 1 dose_Year 8 Group minus Havrix 2 doses_Year 8 Group) of percentage of subjects with anti-HAV antibody concentrations ≥ 15 mIU/mL was to be greater than or equal to the pre-defined clinical non-inferiority limit of -10%; p < 0.0001, Fisher Exact; Difference in seropositivity rate = -23.33, 95% CI 2-sided [-28.78 to -18.29]

6. Secondary Outcome: Number of Subjects With Anti-HAV Antibody Concentrations ≥ 15 mIU/mL at Approximately 10 Years Following Last Administered Havrix Dose - Exploration of Non-inferiority of the 1-dose Schedule Compared to the 2-dose Schedule of Havrix
Description: Subjects are defined as being seropositive if their anti-HAV antibody concentration is equal to or above (≥) 15 mIU/mL.
Time Frame: At approximately 10 years after the last administered vaccine dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group
Number analyzed (Participants) | 299 | 300
Participants | 215 | 289
Statistical Analysis 1: Comparison: Havrix 1 dose_Year 10 Group vs Havrix 2 doses_Year 10 Group; Difference in seropositivity rates for anti-HAV antibody: To demonstrate that 1-dose schedule of Havrix (Havrix 1 dose_Year 10 Group) was non-inferior to the 2-dose schedule of Havrix (Havrix 2 doses_Year 10 Group), in terms of seropositivity rates for anti-HAV antibody, measured by ELISA, approximately 10 years after the administration of the last vaccine dose; Test type: Non-Inferiority — The lower limit of the 2-sided 95% confidence interval (CI) for the difference (Havrix 1 dose_Year 10 Group minus Havrix 2 doses_Year 10 Group) of percentage of subjects with anti-HAV antibody concentrations ≥ 15 mIU/mL was to be greater than or equal to the pre-defined clinical non-inferiority limit of -10%; p < 0.0001, Fisher Exact; Difference in seropositivity rate = -24.43, 95% CI 2-sided [-30.11 to -19.03]

ADVERSE EVENTS:
Time Frame: SAEs: Epoch 001: from Visit at Year 8 (the time of sample collection) up to study conclusion (i.e. during an approximate period of 15 months); Epoch 002: from Visit at Year 10 (the time of sample collection) up to study conclusion (i.e. during an approximate period of 8 months).
Description: Only SAEs related to study procedures were collected during the entire study period.
  There were no other adverse events (AEs) data collected during the entire study period.
Arm/Group | Havrix 1 dose_Year 8 Group | Havrix 2 doses_Year 8 Group | Havrix 1 dose_Year 10 Group | Havrix 2 doses_Year 10 Group
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300 | 0/299 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300 | 0/299 | 0/300
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02712359/SAP_000.pdf
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02712359/Prot_001.pdf